CLINICAL TRIAL: NCT01505114
Title: A Phase II Randomized, Double-Blind, Study of the Safety and Tolerability of Maraviroc (MVC), Maraviroc + Emtricitabine (MVC+FTC), Maraviroc + Tenofovir Disoproxil Fumarate (MVC+TDF), or Tenofovir Disoproxil Fumarate + Emtricitabine (TDF+FTC) For Pre-Exposure Prophylaxis (PrEP) To Prevent HIV Transmission in At-Risk Men Who Have Sex With Men and in At-Risk Women
Brief Title: Evaluating the Safety and Tolerability of Antiretroviral Drug Regimens Used as Pre-Exposure Prophylaxis to Prevent HIV Infection in At-Risk Men Who Have Sex With Men and in At-Risk Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Prevention Trials Network (Network); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HPTN 069/A5305 (NEXT Prep); 11789 (Registry Identifier: DAIDS-ES); HPTN 069/A5305; HPTN 069; HPTN 069/NEXT Prep
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2017-06

CONDITIONS: HIV Infection
Keywords: HIV Prevention; PrEP; Maraviroc
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc; Emtricitabine; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- Arm 1 (Experimental): MVC 300 mg plus FTC placebo and TDF placebo orally once daily
  Interventions: Drug: Maraviroc; Other: Emtricitabine placebo; Other: Tenofovir disoproxil fumarate placebo
- Arm 2 (Experimental): MVC 300 mg plus FTC 200 mg and TDF placebo orally once daily
  Interventions: Drug: Maraviroc; Drug: Emtricitabine; Other: Tenofovir disoproxil fumarate placebo
- Arm 3 (Experimental): MVC 300 mg plus FTC placebo and TDF 300 mg orally once daily
  Interventions: Drug: Maraviroc; Drug: Tenofovir disoproxil fumarate; Other: Emtricitabine placebo
- Arm 4 (Experimental): MVC placebo plus FTC 200 mg and TDF 300 mg orally once daily
  Interventions: Drug: Emtricitabine; Drug: Tenofovir disoproxil fumarate; Other: Maraviroc placebo

INTERVENTIONS:
Drug: Maraviroc — 300-mg tablet, once daily, from Week 0 through Week 48
  Other Names: Selzentry; MVC
  Arms: Arm 1; Arm 2; Arm 3
Drug: Emtricitabine — 200-mg capsule, once daily, from Week 0 through Week 48
  Other Names: Emtriva; FTC
  Arms: Arm 2; Arm 4
Drug: Tenofovir disoproxil fumarate — 300-mg tablet, once daily, from Week 0 through Week 48
  Other Names: Viread; TDF
  Arms: Arm 3; Arm 4
Other: Maraviroc placebo — Once daily from Week 0 through Week 48
  Arms: Arm 4
Other: Emtricitabine placebo — Once daily from Week 0 through Week 48
  Arms: Arm 1; Arm 3
Other: Tenofovir disoproxil fumarate placebo — Once daily from Week 0 through Week 48
  Arms: Arm 1; Arm 2

SUMMARY:
Pre-exposure prophylaxis (PrEP) is a method of preventing HIV infection through the use of antiretroviral (ARV) medications before exposure to HIV. This study will evaluate the safety and tolerability of four ARV regimens in preventing HIV infection in men who have sex with men who may be at risk of getting HIV infection through sex and women who may be at risk of getting HIV infection through sex. The four ARV regimens being evaluated are maraviroc (MVC), MVC plus emtricitabine (FTC), MVC plus tenofovir disoproxil fumarate (TDF), and TDF plus FTC. The MVC-containing arms will be compared to TDF/FTC alone and in combination.

DETAILED DESCRIPTION:
Several clinical trials are currently under way evaluating the safety and efficacy of ARV-based PrEP for preventing HIV infection. In 2010, the results of the first efficacy trial of ARV-based PrEP showed 44% fewer HIV infections among study participants receiving the study drugs (TDF and FTC) than among those receiving placebo. Although these results are promising, concerns about poor adherence, drug resistance, and toxicity prompt further exploration of ARV PrEP regimens. This trial will evaluate the safety and tolerability of PrEP using four ARV regimens in reducing HIV transmission in at-risk men who have sex with men and in at-risk women.

Participants will be randomly assigned to one of four arms: Arm 1, Arm 2, Arm 3, or Arm 4. Arm 1 will receive MVC, FTC placebo, and TDF placebo orally once daily from Week 0 through 48. Arm 2 will receive MVC, FTC, and TDF placebo orally once daily from Week 0 through 48. Arm 3 will receive MVC, FTC placebo, and TDF orally once daily from Week 0 through 48. Participants in Arm 4 will receive MVC placebo, FTC, and TDF orally once daily from Week 0 through 48.

Study visits will occur at enrollment and Weeks 2, 4, 8, 16, 24, 32, 40, 48, and 49. All study visits will include a physical examination, blood collection and storage, and HIV counseling and testing. Select study visits will include adherence counseling, surveys, behavioral assessments (including sexual behavioral assessments), urine collection, and dual-energy x-ray absorptiometry (DXA). Participants will also undergo sexual behavioral assessments randomly 12 to 13 times through Week 48 via short message service (SMS). Some female participants may opt into taking part in an interview at Week 48.

Participants who enroll in this study may also consent to be a part of two subset evaluations as part of this study: the Drug Interaction Subset or the Tissue Subset. Enrollment in these subsets will involve additional study procedures. The Drug Interaction Subset will undergo blood collection before and after a directly observed dose of study drug at the Week 2 visit. Participants in the Tissue Subset will take part in additional study procedures at select visits, including blood collection, hair collection, and rectal tissue and fluid collection (required for men; optional for women). Women involved in the Tissue Subset will also undergo cervical tissue and cervicovaginal fluid collection at select visits.

ELIGIBILITY:
Inclusion Criteria:

* For participants in the men's component of the study, born male. For participants in the women's component of the study, born female.
* 18 years or older at the time of screening
* Willing to provide informed consent for the study
* Able to read at a level required for the study components (e.g., computer-assisted self-interview [CASI] and short message service [SMS], per the judgment of the study investigator)
* For men, a history of receptive or insertive anal intercourse without use of condoms with at least one HIV-infected male partner or male partner of unknown HIV serostatus within 90 days of study entry (provided by self-report)
* For women, a history of vaginal intercourse or receptive anal intercourse without use of condoms with at least one HIV-infected male partner or male partner of unknown HIV serostatus within 90 days of study entry (provided by self-report)
* The following laboratory values must be from specimens obtained within 45 days prior to study enrollment: Nonreactive HIV test results (more information on this criterion can be found in the protocol); hemoglobin (men) greater than 11 g/dL; hemoglobin (women) greater than or equal to 10.5 g/dL; absolute neutrophil count greater than 750 cells/mm^3; platelet count greater than or equal to 100,000/mm^3; for men and women, calculated creatinine clearance greater than or equal to 70 mL/minute using the Cockcroft-Gault equation; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than 3 times the upper limit of normal (ULN); total bilirubin less than 2.5 ULN; urine protein less than 2+; and hepatitis B surface antigen (HBsAg) negative.
* No alcohol or substance use that, in the opinion of the study investigator, would interfere with the conduct of the study (e.g., provided by self-report or found upon medical history and examination or in available medical records)
* No medical condition that, in the opinion of the study investigator, would interfere with the conduct of the study (e.g., provided by self-report or found upon medical history and examination or in available medical records)
* Willing to undergo all required study procedures (including sexual assessment by CASI, use of the drug monitoring device, and SMS [i.e., texting])
* For all women participants: If of reproductive potential (defined as girls who have reached menarche and pre-menopausal women who have not had a sterilization procedure per self-report (e.g., hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy), must have a negative serum or urine pregnancy test performed within 48 hours before initiating the protocol-specified medication(s). More information on this criterion can be found in the protocol.
* For all women participants: If participating in sexual activity that could lead to pregnancy, must agree to use a form of contraception from the following list during the trial and for 30 days after stopping the study medication: condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, IUD, or hormone-base contraceptive.

Inclusion Criteria for the Tissue Subset:

* For men and women participating in the rectal component, willing to abstain from receptive anal intercourse and practices involving insertion of anything in the rectum (drug, enema, penis, or sex toy) for 3 days prior to rectal biopsy and for 7 days post-biopsy, to minimize risk of HIV-1 infection and bleeding complications after each procedure
* For women participating in the vaginal component, willing to abstain from vaginal intercourse and practices involving insertion of anything in the vagina (drug, douche, penis, or sex toy) for 3 days prior to cervical biopsy and for 7 days post-biopsy, to minimize risk of HIV-1 infection and bleeding complications after each procedure
* For women only, per participant report at screening, usual menstrual cycle with at least 21 days between menses (does not apply to participants who report using a progestin-only method of contraception at screening, e.g., Depo-Provera)
* For women, satisfactory Pap results in the 12 calendar months prior to enrollment consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009), or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result per American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines in the 12 calendar months prior to enrollment. If there is no document of satisfactory Pap results, the participant should be offered to have the test performed by the site prior to the enrollment visit. If they refuse, they are not eligible.

Exclusion Criteria:

* One or more reactive HIV test results at screening or enrollment, even if HIV infection is not confirmed
* Coenrollment in any other HIV interventional research study (provided by self-report or other available documentation) or prior enrollment and receipt of active arm (i.e., NOT a placebo) of an HIV vaccine trial (provided by available documentation)
* Use of ARV therapy (e.g., for post-exposure prophylaxis [PEP] or PrEP) in the 90 days prior to study entry
* Prior history of a gastrectomy, colostomy, ileostomy, or any other procedure altering the gastrointestinal tract or drug absorption (provided by self-report or obtained from medical history or records)
* Receipt of prohibited medications as described in the study drug package inserts or listed in the Study-Specific Populations (SSP) Manual (provided by self-report or obtained from medical history or medical records)
* Ongoing intravenous drug use: episodic use or any use in the past 90 days (as assessed by the study investigator)
* Known medical history of allergy to soy (soya or soybeans) or peanuts
* Weight exceeding 300 pounds (exceeds weight limit of DXA scanners)
* For women, pregnancy or currently breastfeeding

Exclusion Criteria for the Tissue Subset:

For Men and Women:

* The following applies to men, and only to women who opt for rectal sampling: Abnormalities of the colorectal mucosa or significant colorectal symptom(s), which in the opinion of the study investigator represent a contraindication to biopsy (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of symptomatic external hemorrhoids)
* Per participant report at screening, anticipated use and/or unwillingness to abstain from the following medications during the period of study participation: Heparin, including Lovenox®, Warfarin, Plavix® (clopidogrel bisulfate), or any other drugs that are associated with increased risk of bleeding following biopsy procedures in the opinion of the study investigator
* The following applies to men, and only to women who opt for rectal sampling: Per participant report at screening, anticipated use and/or unwillingness to abstain from rectally administered medications (including over-the-counter products) for 3 days prior to rectal biopsies and for 7 days after biopsies
* Per participant report at screening, anticipated use and/or unwillingness to abstain from the following medications for a period of 10 days before a biopsy procedure: aspirin (daily use of low-dose aspirin [no more than 81 mg] is allowed at the discretion of the Investigator of Record) or non-steroidal anti-inflammatory drugs (NSAIDS)
* Abnormal laboratory results for coagulation tests that may indicate an increased risk of bleeding (in the opinion of the investigators)
* Active untreated syphilis, gonorrhea, or chlamydia infection

For Women Only:

* Carcinoma in situ of the cervix or invasive cervical cancer. Abnormalities of the vaginal mucosa or significant vaginal symptom(s), which in the opinion of the study investigator represent a contraindication to biopsy (including but not limited to presence of any unresolved injury, and infectious or inflammatory condition of the local mucosa).
* Hysterectomy
* Per participant report at screening, anticipated use and/or unwillingness to abstain from vaginally administered medications (including over-the-counter products) and vaginal douching for 3 days prior to cervical biopsies and for 7 days after biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy M. Gulick, MD, MPH, Study Chair — Weill Medical College of Cornell University
Locations (13):
- United States (12):
  - UCLA CARE Center CRS, Los Angeles, California
  - Bridge HIV CRS, San Francisco, California
  - George Washington Univ. CRS, Washington D.C., District of Columbia
  - Johns Hopkins University CRS, Baltimore, Maryland
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Brown KC, Patterson KB, Malone SA, Shaheen NJ, Prince HM, Dumond JB, Spacek MB, Heidt PE, Cohen MS, Kashuba AD. Single and multiple dose pharmacokinetics of maraviroc in saliva, semen, and rectal tissue of healthy HIV-negative men. J Infect Dis. 2011 May 15;203(10):1484-90. doi: 10.1093/infdis/jir059. PMID 21502084
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Derived] Kapadia SN, Wu C, Mayer KH, Wilkin TJ, Amico KR, Landovitz RJ, Andrade A, Chen YQ, Chege W, McCauley M, Gulick RM, Schackman BR. No change in health-related quality of life for at-risk U.S. women and men starting HIV pre-exposure prophylaxis (PrEP): Findings from HPTN 069/ACTG A5305. PLoS One. 2018 Dec 26;13(12):e0206577. doi: 10.1371/journal.pone.0206577. eCollection 2018. PMID 30586364
- [Derived] Gulick RM, Wilkin TJ, Chen YQ, Landovitz RJ, Amico KR, Young AM, Richardson P, Marzinke MA, Hendrix CW, Eshleman SH, McGowan I, Cottle LM, Andrade A, Marcus C, Klingman KL, Chege W, Rinehart AR, Rooney JF, Andrew P, Salata RA, Siegel M, Manabe YC, Frank I, Ho K, Santana J, Stekler JD, Swaminathan S, McCauley M, Hodder S, Mayer KH. Safety and Tolerability of Maraviroc-Containing Regimens to Prevent HIV Infection in Women: A Phase 2 Randomized Trial. Ann Intern Med. 2017 Sep 19;167(6):384-393. doi: 10.7326/M17-0520. Epub 2017 Aug 22. PMID 28828489
- [Derived] Gulick RM, Wilkin TJ, Chen YQ, Landovitz RJ, Amico KR, Young AM, Richardson P, Marzinke MA, Hendrix CW, Eshleman SH, McGowan I, Cottle LM, Andrade A, Marcus C, Klingman KL, Chege W, Rinehart AR, Rooney JF, Andrew P, Salata RA, Magnus M, Farley JE, Liu A, Frank I, Ho K, Santana J, Stekler JD, McCauley M, Mayer KH. Phase 2 Study of the Safety and Tolerability of Maraviroc-Containing Regimens to Prevent HIV Infection in Men Who Have Sex With Men (HPTN 069/ACTG A5305). J Infect Dis. 2017 Jan 15;215(2):238-246. doi: 10.1093/infdis/jiw525. PMID 27811319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started the enrollment in June 2012. Accrual will occur in a staggered fashion, with men beginning first and women beginning several months later. Accrual for the men will occur over approximately 9 months, and accrual for the women will require approximately 9 months.
Pre-assignment Details: Exclusion--reactive HIV test results;Co-enrollment in any other HIV interventional research study; Use of ARV therapy; Prior history of any procedure altering the gastrointestinal tract or drug absorption; Receipt of prohibited medications; Known allergy to soy/peanuts; Weight>300 lbs;
Groups:
- MVC Only: MVC 300 mg plus FTC placebo and TDF placebo orally once daily
  Maraviroc: 300-mg tablet, once daily, from Week 0 through Week 48
  Emtricitabine placebo: Once daily from Week 0 through Week 48
  Tenofovir disoproxil fumarate placebo: Once daily from Week 0 through Week 48
- MVC + FTC: MVC 300 mg plus FTC 200 mg and TDF placebo orally once daily
  Maraviroc: 300-mg tablet, once daily, from Week 0 through Week 48
  Emtricitabine: 200-mg capsule, once daily, from Week 0 through Week 48
  Tenofovir disoproxil fumarate placebo: Once daily from Week 0 through Week 48
- MVC + TDF: MVC 300 mg plus FTC placebo and TDF 300 mg orally once daily
  Maraviroc: 300-mg tablet, once daily, from Week 0 through Week 48
  Tenofovir disoproxil fumarate: 300-mg tablet, once daily, from Week 0 through Week 48
  Emtricitabine placebo: Once daily from Week 0 through Week 48
- TDF + FTC: MVC placebo plus FTC 200 mg and TDF 300 mg orally once daily
  Emtricitabine: 200-mg capsule, once daily, from Week 0 through Week 48
  Tenofovir disoproxil fumarate: 300-mg tablet, once daily, from Week 0 through Week 48
  Maraviroc placebo: Once daily from Week 0 through Week 48
Period: Overall Study
Arm/Group | MVC Only | MVC + FTC | MVC + TDF | TDF + FTC
Started | 148 | 148 | 147 | 151
Completed | 123 | 135 | 129 | 128
Not Completed | 25 | 13 | 18 | 23
Not completed — Withdrawal by Subject | 5 | 4 | 4 | 7
Not completed — Death | 1 | 0 | 0 | 1
Not completed — unable to adhere to visit schedule | 3 | 2 | 3 | 3
Not completed — Lost to Follow-up | 11 | 5 | 8 | 7
Not completed — relocated | 4 | 2 | 2 | 3
Not completed — inadvertent enrollment due to peanut all | 0 | 0 | 0 | 1
Not completed — staff safety concerns | 0 | 0 | 0 | 1
Not completed — investigator decision | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 147 | 151 | 148 | 148 | 594
Age, Continuous [Median (Full Range); unit: years] — Population: analysis for men
  years
    number analyzed (Participants) | 101 | 106 | 99 | 100 | 406
    (all) | 30 [18 to 65] | 29.5 [18 to 62] | 30 [18 to 70] | 31 [18 to 60] | 30 [18 to 70]
Age, Continuous [Median (Full Range); unit: years] — Population: Analysis for women
  years
    Women: number analyzed (Participants) | 46 | 45 | 49 | 48 | 188
    Women | 40 [18 to 61] | 36 [19 to 57] | 37 [22 to 60] | 37 [18 to 60] | 36 [18 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 49 | 48 | 188
  Male | 101 | 106 | 99 | 100 | 406
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 4 | 6 | 2 | 5 | 17
  Asian | 6 | 1 | 5 | 5 | 17
  Black or African | 61 | 64 | 62 | 51 | 238
  Native Hawaiian or Pacific Islander | 1 | 2 | 1 | 3 | 7
  White | 73 | 80 | 72 | 78 | 303
  Other | 15 | 14 | 10 | 16 | 55
education [Count of Participants; unit: Participants]
  8th Grade or Less | 1 | 3 | 0 | 1 | 5
  Some High School | 10 | 7 | 6 | 9 | 32
  High School Graduate or Equivalent | 35 | 27 | 25 | 27 | 114
  Vocational/Trade/Technical School | 3 | 7 | 7 | 6 | 23
  Some College or 2 Year Degree | 51 | 43 | 57 | 55 | 206
  Finished College | 37 | 40 | 36 | 40 | 153
  masters or other advanced degree | 10 | 24 | 17 | 10 | 61
Marital Status [Count of Participants; unit: Participants]
  Married/Civil Union/Legal Partnership | 8 | 9 | 7 | 14 | 38
  Living with Primary Partner | 25 | 21 | 25 | 21 | 92
  Not Living with Primary Partner | 12 | 17 | 19 | 14 | 62
  Single/Divorced/Widowed | 102 | 103 | 96 | 98 | 399
  Other | 0 | 1 | 1 | 1 | 3
Employment Status [Count of Participants; unit: Participants]
  Full-time Employment | 56 | 68 | 59 | 74 | 257
  Part-time Employment | 38 | 35 | 36 | 25 | 134
  Not Employed | 53 | 48 | 52 | 49 | 202

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Grade 3 or Higher Adverse Events (AEs)
Description: participants had Occurrence of Grade 3 or higher adverse events (AEs)
Time Frame: Through Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 147 | 151 | 148 | 148
Participants | 18 | 24 | 20 | 28

ADVERSE EVENTS:
Time Frame: 49 weeks
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
All-Cause Mortality (participants affected / at risk) | 0/147 | 1/151 | 1/148 | 0/148
Serious Adverse Events (participants affected / at risk) | 10/147 | 5/151 | 4/148 | 11/148
Other Adverse Events (participants affected / at risk) | 78/147 | 86/151 | 84/148 | 91/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=147) | Arm 2 (N=151) | Arm 3 (N=148) | Arm 4 (N=148)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital anomaly in offspring (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chikungunya virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion late (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=147) | Arm 2 (N=151) | Arm 3 (N=148) | Arm 4 (N=148)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (5)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anogenital dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Anorectal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 13 (13) | 6 (6) | 3 (3) | 8 (11)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Gingival recession (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 6 (6) | 2 (2) | 5 (6)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fat tissue increased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 2 (2) | 3 (3) | 1 (1) | 4 (4)
Malaise (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Allergy to animal (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (2)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal chlamydia infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Anal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cellulitis of male external genital organ (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chikungunya virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 4 (4) | 4 (6) | 1 (1) | 5 (5)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatophytosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Endometritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 6 (6) | 2 (2) | 4 (4)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (5)
Genitourinary tract gonococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gonorrhoea (Infections and infestations) | 3 (3) | 4 (4) | 2 (2) | 3 (3)
Herpes simplex (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infected bite (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 3 (4) | 2 (2) | 5 (5)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (3)
Oral pustule (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 4 (4) | 0 (0) | 3 (3) | 3 (3)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otitis media bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Papilloma viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngeal chlamydia infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis bacterial (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 5 (5) | 6 (6) | 2 (3)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Primary syphilis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Proctitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctitis chlamydial (Infections and infestations) | 10 (11) | 2 (3) | 3 (4) | 5 (5)
Proctitis gonococcal (Infections and infestations) | 4 (4) | 5 (5) | 5 (5) | 3 (3)
Proctitis herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Secondary syphilis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 5 (6) | 1 (1) | 2 (2) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Syphilis (Infections and infestations) | 3 (3) | 2 (2) | 5 (5) | 3 (3)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 9 (10) | 6 (7) | 9 (9)
Urethritis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Urethritis chlamydial (Infections and infestations) | 1 (2) | 6 (8) | 2 (2) | 3 (3)
Urethritis gonococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (6) | 6 (8) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 8 (8) | 11 (12) | 6 (6) | 3 (3)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic iritis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 8 (10) | 5 (6) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 7 (8) | 3 (3) | 4 (5)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 3 (3) | 2 (3) | 5 (8)
Blood cholesterol increased (Investigations) | 1 (1) | 3 (3) | 6 (6) | 6 (6)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Blood glucose decreased (Investigations) | 3 (3) | 2 (3) | 8 (9) | 3 (3)
Blood glucose increased (Investigations) | 3 (6) | 5 (9) | 3 (3) | 7 (10)
Blood phosphorus decreased (Investigations) | 9 (13) | 13 (13) | 11 (13) | 12 (17)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Carbon dioxide decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine urine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 2 (3) | 2 (2) | 0 (0) | 3 (4)
Lipids increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 4 (5) | 6 (7) | 6 (6)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (4) | 4 (6) | 2 (2) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (5)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (3) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 4 (7) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 12 (21) | 15 (23) | 13 (19) | 7 (10)
Lactose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4) | 5 (5) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (9) | 8 (8) | 6 (7) | 6 (7)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Motor dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (9) | 6 (6) | 5 (6) | 2 (3)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 3 (5) | 2 (2) | 1 (1)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Substance abuse (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thinking abnormal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tobacco withdrawal symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3) | 3 (3) | 2 (3) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 8 (9) | 3 (3) | 4 (4) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethral discharge (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital lesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penile discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne cystic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dandruff (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hyperaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study abstracts and publications are subject to HPTN Publication and Public Information Policies and Clinical Trial Agreements between NIAID (DAIDS) and company collaborators. The publication or other disclosure can be delayed for up to thirty additional business days for manuscripts & five business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.